CLINICAL TRIAL: NCT07372339
Title: Comparison of Breast Sensory Recovery Between Conventional and Endoscopic Nipple-Sparing Mastectomy Combined With Prepectoral Implant Reconstruction：an Open-label, Multicentre, Randomised, Controlled Trial
Brief Title: Comparison of Breast Sensory Recovery Between Conventional and Endoscopic Nipple-Sparing Mastectomy Combined With Prepectoral Implant Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJMU-BC11
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional nipple-sparing mastectomy group (Experimental)
  Interventions: Procedure: Conventional nipple-sparing mastectomy combined with prepectoral implant reconstruction
- Endoscopic nipple-sparing mastectomy group (Active Comparator)
  Interventions: Procedure: Endoscopic nipple-sparing mastectomy combined with prepectoral implant reconstruction

INTERVENTIONS:
Procedure: Conventional nipple-sparing mastectomy combined with prepectoral implant reconstruction — This procedure is a traditional surgical approach involving a skin incision made on the breast surface. Under direct visualization, the breast glandular tissue is excised while preserving the nipple-areola complex, followed by a reconstructive surgery with implant placement in the prepectoral plane.
  Arms: Conventional nipple-sparing mastectomy group
Procedure: Endoscopic nipple-sparing mastectomy combined with prepectoral implant reconstruction — This minimally invasive procedure is performed through small, concealed incisions in the axilla. Utilizing endoscopic instruments and an imaging system, the breast glandular tissue is resected under video monitoring, followed by reconstructive surgery with implant placement in the prepectoral plane.
  Arms: Endoscopic nipple-sparing mastectomy group

SUMMARY:
This clinical trial aims to determine whether conventional surgery or endoscopic surgery results in better recovery of breast skin sensation in women with early-stage breast cancer undergoing nipple-sparing mastectomy with prepectoral implant reconstruction. Furthermore, the study will compare the safety, aesthetic outcomes, and quality of life associated with the two surgical approaches. The study seeks to address the following primary research questions:

Does conventional surgery lead to superior recovery of breast skin sensation at 6 months postoperatively compared with endoscopic surgery?

What are the differences between the two surgical approaches in terms of complication rates, aesthetic outcomes, and patient-reported quality of life?

Researchers will compare conventional nipple-sparing mastectomy with endoscopic nipple-sparing mastectomy to determine which procedure better preserves postoperative breast sensation.

Participants will:

Be randomly assigned to undergo either conventional or endoscopic surgery.

Have breast skin sensation measured preoperatively and at multiple postoperative follow-up visits using a standardized assessment tool.

Complete validated questionnaires regarding breast satisfaction and quality of life preoperatively and during multiple follow-up visits.

Attend scheduled follow-up visits to monitor for complications and to evaluate the long-term appearance and health of the reconstructed breast.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 to 70 years.
2. Unilateral breast cancer confirmed by preoperative pathology.
3. Scheduled to undergo nipple-sparing mastectomy (NSM) with immediate prepectoral implant-based breast reconstruction.
4. Invasive carcinoma with a maximum tumor diameter ≤ 5 cm, or ductal carcinoma in situ (DCIS).
5. Preoperative imaging assessment confirms a distance of ≥ 1 cm between the lesion and the nipple-areola complex (NAC).
6. No clinical, radiological, or pathological evidence of tumor invasion into the NAC, skin, or pectoralis major muscle. The tumor must be confined within the glandular tissue.
7. No evidence of distant metastasis (M0).
8. Clinically node-negative (cN0) as assessed by preoperative examination.
9. No history of neoadjuvant chemotherapy or radiotherapy prior to surgery.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Willing and able to understand the study procedures, provide written informed consent, demonstrate good compliance, and agree to participate in follow-up evaluations.
12. The principal surgeon must have experience in performing at least 30 cases of NSM combined with implant-based reconstruction.

Exclusion Criteria:

1. Diagnosis of Paget's disease of the breast, recurrent breast cancer, or a history of prior thoracic radiation therapy.
2. Evidence of tumor invasion into the skin (including inflammatory breast cancer), nipple-areola complex, or pectoralis major muscle.
3. Pregnancy or lactation at the time of enrollment.
4. Requirement for re-excision following a prior breast lump biopsy, or a history of any previous breast surgery (including but not limited to augmentation mammoplasty, breast reduction, lumpectomy, etc.).
5. Breast size exceeding a D-cup.
6. Body mass index (BMI) > 30 kg/m².
7. Grade III ptosis (severe breast drooping where the nipple is positioned below the inframammary fold).
8. Pre-existing nipple-areolar complex deformities (e.g., nipple inversion, areolar hypoplasia), active skin conditions of the breast (e.g., eczema, dermatitis, infection, ulceration), or significant scarring compromising the surgical site.
9. Severe systemic comorbidities (e.g., immunosuppression, uncontrolled diabetes mellitus, severe cardiopulmonary dysfunction, coagulopathy or bleeding diathesis, contraindications to general anesthesia).
10. Known hypersensitivity or allergy to silicone gel implants, or to anesthetic agents/antibiotics used perioperatively.
11. Pre-existing neurological disorders (e.g., diabetic peripheral neuropathy, Parkinson's disease, polyneuritis, spinal cord injury) or chronic use of medications known to affect neurological/sensory function (e.g., antidepressants, antiepileptics).
12. Current heavy smoking (>20 cigarettes per day).
13. Current alcohol abuse or substance addiction.
14. Concurrent or history of other active malignancies
15. Anticipated poor compliance with follow-up protocols or inability to complete scheduled postoperative evaluations.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Average breast sensory thresholds at 6 months post breast reconstruction as measured by Semmes-Weinstein Monofilaments | 6 months
  Differences in the mean skin sensory thresholds (measured by Semmes-Weinstein monofilaments across nine breast regions) between the conventional and endoscopic surgery groups were observed at 6 months after breast reconstruction.

SECONDARY OUTCOMES:
Number of participants with postoperative complications as assessed by Clavien-Dindo Classification System within 1 year after surgery | within 1 year
  Complications (e.g., hematoma, infection, flap necrosis) will be recorded and graded according to the Clavien-Dindo Classification System. The outcome is the count (and percentage) of participants experiencing at least one complication within the first postoperative year. These events are assessed at scheduled follow-up visits at 1, 3, 6, and 12 months.
Patient-reported quality of life as measured by Breast-Q reconstruction module | 6 months and 1 year
  The Breast-Q reconstruction module assesses multiple domains, including psychosocial well-being, sexual well-being, physical well-being (of the chest and upper body), and satisfaction with breasts. All scores are transformed to a 0-100 scale.
Physician-assessed breast aesthetic score using a 5-point Likert scale | 6 months and 1 year
  Independent surgeons will rate five specific domains (volume, shape, symmetry, scar, NAC) on a 5-point Likert scale (1=very dissatisfied to 5=very satisfied) using blinded photographs. The mean score for each domain and the composite mean score will be compared between groups.
Patient-reported quality of life as assessed by E0RTC QLQ-C30 | 6 months and 1 year
  Patient-reported quality of life measured by E0RTC QLQ-C30, consists of 30 items grouped into functional scales, symptom scales and single items, global health status scale. Responses for most items are recorded on a 4-point Likert scale (1="Not at all" to 4="Very much"). The two Global Health Status items use a 7-point linear analogue scale (1="Very poor" to 7="Excellent"). Raw scores are linearly transformed to a standardized score ranging from 0 to 100 for each scale. For the functional scales and the global health status scale: a higher score indicates a better level of functioning or quality of life. For the symptom scales / single Items: a higher score indicates a greater severity of symptoms or problems.
Long-term breast skin sensation threshold as measured by Semmes-Weinstein Monofilaments | Annually up to 10 years
  The mean pressure threshold, measured in grams using the Semmes-Weinstein monofilament test across nine standardized breast regions, will be compared between the conventional surgery group and the endoscopic surgery group after nipple-sparing mastectomy with prepectoral implant reconstruction for a long time.
Number of participants with postoperative complications as assessed by Clavien-Dindo Classification System after surgery in the long term. | Annually up to 10 years
  Number of participants with postoperative complications assessed by Clavien-Dindo Classification System will be compared between two groups annually in the long term.
Long-term physician-assessed breast aesthetic score | Annually up to 10 years
  Independent surgeons will rate five specific domains (volume, shape, symmetry, scar, NAC) on a 5-point Likert scale (1=very dissatisfied to 5=very satisfied) using blinded photographs. The mean score will be compared between groups at annual follow-ups.
Long-term patient-reported quality of life as measured by Breast-Q reconstruction module | Annually up to 10 years
  The Breast-Q reconstruction module assesses multiple domains, including psychosocial well-being, sexual well-being, physical well-being (of the chest and upper body), and satisfaction with breasts. All scores are transformed to a 0-100 scale. The mean score will be compared between groups at annual follow-ups.
Long-term patient-reported quality of life as assessed by EORTC-QLQ-C30 | Annually up to 10 years
  Long-term patient-reported quality of life measured by E0RTC QLQ-C30, consists of 30 items grouped into functional scales, symptom scales and single items, global health status scale. Responses for most items are recorded on a 4-point Likert scale (1="Not at all" to 4="Very much"). The two Global Health Status items use a 7-point linear analogue scale (1="Very poor" to 7="Excellent"). Raw scores are linearly transformed to a standardized score ranging from 0 to 100 for each scale. For the functional scales and the global health status scale: a higher score indicates a better level of functioning or quality of life. For the symptom scales / single Items: a higher score indicates a greater severity of symptoms or problems.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JH, Ryu JM, Bae SJ, Ko BS, Choi JE, Kim KS, Cha C, Choi YJ, Lee HY, Nam SE, Kim Z, Kang YJ, Lee MH, Lee JE, Park E, Shin HJ, Kim MK, Choi HJ, Kwon SU, Son NH, Park HS, Lee J; Korea Robot-endoscopy Minimal Access Breast Surgery Study Group. Minimal Access vs Conventional Nipple-Sparing Mastectomy. JAMA Surg. 2024 Oct 1;159(10):1177-1186. doi: 10.1001/jamasurg.2024.2977. PMID 39141399
- [Background] Hammond JB, Kandi LA, Armstrong VL, Kosiorek HE, Rebecca AM, Casey WJ 3rd, Kruger EA, Cronin PA, Pockaj BA, Teven CM. Long-term breast and nipple sensation after nipple-sparing mastectomy with implant reconstruction: Relevance to physical, psychosocial, and sexual well-being. J Plast Reconstr Aesthet Surg. 2022 Sep;75(9):2914-2919. doi: 10.1016/j.bjps.2022.06.034. Epub 2022 Jun 20. PMID 35915018
- [Background] Lai HW, Chang YL, Chandrachamnong K, See MH, Huang HI, Lin SL, Fang DY, Chen ST, Chen DR, Mok CW, Cheng FT. Factors associated with alteration of nipple or skin sensation and impact of duration of time following nipple-sparing mastectomy (NSM): an analysis of 460 cases with comparison of conventional versus endoscopic- or robotic-assisted NSM. World J Surg Oncol. 2023 Jul 26;21(1):222. doi: 10.1186/s12957-023-03107-5. PMID 37491239
- [Background] Zhou J, Xie Y, Liang F, Feng Y, Yang H, Qiu M, Zhang Q, Chung K, Dai H, Liu Y, Liang P, Du Z. A novel technique of reverse-sequence endoscopic nipple-sparing mastectomy with direct-to-implant breast reconstruction: medium-term oncological safety outcomes and feasibility of 24-h discharge for breast cancer patients. Int J Surg. 2024 Apr 1;110(4):2243-2252. doi: 10.1097/JS9.0000000000001134. PMID 38348883
- [Background] Seth AK, Sisco M. Prepectoral Breast Reconstruction. Plast Reconstr Surg. 2025 Jan 1;155(1):213e-227e. doi: 10.1097/PRS.0000000000011737. Epub 2024 Dec 16. PMID 39700251